CLINICAL TRIAL: NCT05758506
Title: Developing a Screening Tool for Primary Immunodeficiency Disease (PID) in Pakistan
Status: Completed | Type: Observational
Sponsor: PATH (Other)
Responsible Party: Principal Investigator, Megan Parker, Senior Research Research Officer, Diagnostics, PATH
Other Study IDs: 1840225
Record Dates: First submitted 2022-11-10; First posted 2023-03-07 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Primary Immunodeficiency Diseases
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pediatric PID patients (prospective): Prospective, age-matched, healthy patients
  Interventions: Device: Primary Immunodeficiency (PID) Rapid Diagnostic Test (RDT)
- Pediatric PID patients (recontacted from registry)
  Interventions: Device: Primary Immunodeficiency (PID) Rapid Diagnostic Test (RDT)
- Prospective, age-matched, healthy patients
  Interventions: Device: Primary Immunodeficiency (PID) Rapid Diagnostic Test (RDT)

INTERVENTIONS:
Device: Primary Immunodeficiency (PID) Rapid Diagnostic Test (RDT) — We are evaluating the accuracy of a new rapid diagnostic screening test. There is no medical intervention with the participants in this study.

SUMMARY:
Case-control diagnostic accuracy study with 130 potential pediatric PID+ (primary immunodeficiency) patients, and 100 age-matched, healthy controls (PID-). The potential PID+ participants will be recruited prospectively through 9 hospitals in Sindh and Punjab states or contacted via the PID surveillance registry developed by AKU Hospital's Polio Excretion in PID study to identify children with primary antibody deficiency (PAD+: a type of PID+); healthy, age-matched PID-participants will be recruited by snowball sampling. At the point of care, health care workers (HCWs) will collect capillary blood samples (0.1mL) to run the PID rapid screening test and reader on potential PID+ participants (identified by exhibiting >2 of the Jeffrey Modell warning signs) and healthy, age-matched controls. All pediatric study participants will be sent to the hospital lab to have a confirmatory immunology panel (see 4.4.1 Diagnosing PID for the battery of tests) run on a serum/plasma sample to confirm their PID diagnosis (PID+/PAD-, PID+/PAD+, PID-); a 1.5uL aliquot of serum/plasma will simultaneously be used to run a PID rapid screening test by a laboratory technician (LT). HCWs and LTs will be blinded to true PID status. Blood and serum PID rapid screening test results will be compared to the confirmatory immunology panel to determine diagnostic accuracy. All clinical management of study participants will follow the standard of care for PID in Pakistan and will be based upon the immunology panel result. The HCWs and LTs administering the tests will be trained prior to the diagnostic accuracy test (see Objectives below) and will provide feedback on the tool post-training and post-use to assess usability, acceptability, and feasibility of integrating the test and digital reader into tertiary hospitals for the purpose of improved national PID surveillance, improved PID patient care, and polio eradication in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3 months to 15 years

  * Presents for care at 1 of 9tertiary hospitals participating in the study
  * Potential PID+ (Case): Child is identified by HCW to have >2 Jeffrey Model warning signs of PID. [Note: Upon immunology panel testing, this group will be separated into three categories: PID-, PID+, and PID+/PAD+ meaning they have 1 of 5 relevant primary antibody deficiencies (PAD+)].
  * PID-(Control): Child is identified (by snowball sampling) as being in good health, and having the same age (within 12 months) as another child who produced a PID+ result.
  * Caregiver consents to participate in the study and provides informed consent. If their children are 10 years of age or older, that child must also give assent.

Exclusion Criteria:

* Aged less than 3 months or greater than 15 years of age

  * Caregiver does not consent to participate, or child >10years does not give assent to participate.
  * Having received IVIG in the past 90 days

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: - 130 potential PID patients with (5 relevant PIDs: PADs) within Sindh and Punjab states V1.0, 6 Jan 2022
  • 100 healthy, age-matched children within Sindh and Punjab state
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 8 month
  Estimates of diagnostic accuracy characteristics with 95% confidence intervals (sensitivity, specificity, PPV, NPV) of the PID screening test for relevant PIDs in a Pakistani population of both PID+ children and PID- age-matched healthy controls
Determine usability, acceptability, feasibility of integrating PID test and digital reader into tertiary hospitals for improved patient care | 8 months
  Estimates of user effectiveness, efficacy, satisfaction, learnability, and feasibility among trained health care workers (HCWs) and laboratory technicians (LTs) will be evaluated using observation checklists and surveys. The observation checklist will evaluate the ability to administer the test, read the test results accurately after the appropriate amount of waiting time, record the result in the digital reader app, operate the digital app to read a photograph of the test result, and their ease of performing these tasks. This methodology adheres to ISO 9241-210 on human-centered design principles in usability testing.

SECONDARY OUTCOMES:
Effectiveness - agreement between the PID screening test readouts (#1, #2) with each other, the digital reading, a PATH expert panel, and the local PID standard of care immunology tests. | 8 months
  Percent (%) agreement between each of the PID screening test results, digital app result, expert panel, and immunology panel.
Effectiveness | 8 months
  Percent (%) agreement in PID screening test results between capillary whole blood samples and serum samples.
Understandability of diagnostic instruction | 8 months
  Percent of trained end users who can accurately comprehend the material presented in the training course curriculum and the IFU.
Usability of screening test result outputs | 8 months
  Percent of trained end users who can accurately interpret the investigational device result output.
Usability for facilitators | 8 months
  Percent of stakeholders who would use the test, lists of barriers and facilitators cited for Pakistani context.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The data generated by this study will inform decisions regarding product development and commercialization of the BioSure PID rapid screening test and digital reader. The data collected in this evaluation may be used to support regulatory approval of the test. The study will generate valuable data on the performance of this novel test in comparison to that of the Jeffrey Modell warning signs and the immunology panel enabling informed decision-making regarding recommendation of new highly sensitive POC tools for PID. Data will be shared with study partners and the test developers. This may include de-identified, individual-level data.
Supporting Information: Study Protocol